CLINICAL TRIAL: NCT05689008
Title: Efficacy and Safety of Umbilical Cord Mesenchymal Stem Cells in the Treatment of Severe and Critical COVID-19 With Refractory Hypoxia
Brief Title: UC-MSCs in the Treatment of Severe and Critical COVID-19 Patients With Refractory Hypoxia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai East Hospital (Other)
Collaborators: Sir Run Run Shaw Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DFSC-2023(CR)-01
Record Dates: First submitted 2023-01-17; First posted 2023-01-18 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Mesenchymal Stem Cell; COVID-19 Pneumonia
Keywords: umbilical cord mesenchymal stem cells; covid-19 pneumonia; refractory hypoxia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (No Intervention): Participants will receive standard therapy, including oxygen therapy，glucocorticoid and other antiinflammatory drugs and supportive treatments according the ninth edition of Chinese guidelines for the treatment of COVID-19 infection.
- UC-MSCs treatment (Experimental): Participants will receive two doses of UC-MSCs instillation at the first and fourth day after the assignment on the basis of standard treatment.
  Interventions: Biological: UC-MSCs treatment

INTERVENTIONS:
Biological: UC-MSCs treatment — Participants will receive two doses of UC-MSCs treatment, each dose will contain 1*10^6 cells/kg suspended in 100 ml albumin solution.
  Arms: UC-MSCs treatment

SUMMARY:
The goal of this randomized, controlled, open-labeled interventional clinical trial is to test the efficacy and safety of umbilical cord mesenchymal stem cells (UC- MSCs) in the treatment of severe and critical COVID-19 patients with refractory hypoxia even after sufficient standard treatment according to the tenth edition of Chinese guidelines for COVID-19 infection. The main questions it aims to answer are: 1. The efficacy of UC-MSCs in the treatment of severe and critical COVID-19 patients with refractory hypoxia. 2. The safety of UC-MSCs in the treatment of severe and critical COVID-19 patients. 3. The potential immune mechanisms of UC- MSCs in the treatment of severe and critical COVID-19 patients. Participants will receive standard therapy, or the UC-MSCs treatment. For the standard treatment, it will be conducted according the 10th edition of Chinese guidelines for severe or critical COVID-19 infection. For UC-MSCs treatment, participants will be given UC-MSCs instillation at the first and fourth day after assignment. Blood examples will be taken at indicated time for arterial blood gas analysis and other tests. And participants should also objectively report their symptoms change and other information related to the treatment as listed the research protocol.

ELIGIBILITY:
Inclusion Criteria:

* The age ranges from 18 to85 (inclusive), regardless of gender.
* Patients who still have refractory hypoxia after sufficient standard treatment for severe and critical COVID-19 pneumonia following the suggestion of the Chinese diagnostic criteria for COVID-19 pneumonia in the Diagnosis and Treatment Plan for COVID-19 Pneumonia (Tentative tenth Edition).
* 20kg/m2≤body mass index(BMI)≤30 kg/m2.
* Volunteer to participate in this clinical study and sign the written informed consent

Exclusion Criteria:

* Those who are using immunosuppressive drugs or long-term immunosuppressive drugs after organ transplantation.
* T lymphocyte abnormality (allogeneic may be considered, depending on clinical opinion), HIV positive.
* Highly allergic or have a history of severe allergy, especially Interleukin-2 allergy.
* Pregnant and lactating women.
* Patients with severe autoimmune disease history; Allergies to all biological reagents in this treatment, such as Interleukin-2.
* Patients with serious complications, including chronic cardiac insufficiency (NYHA cardiac function grading assessment of cardiac function grade III - IV), chronic renal insufficiency (CKD stage 3 and above); Chronic liver insufficiency (Child-Pugh score>7); Patients with malignant tumors.
* Patients with pulmonary embolism or acute coronary syndrome.
* Patients with severe organ dysfunction caused by other diseases.
* There are other situations that the researcher thinks are not suitable to participate in this clinical study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-10 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
Oxygenation index | Change from baseline Oxygenation index (PaO2/FiO2) at 1,3,7,14,28 (or before the day of discharge if participants discharge within 28 days) days after the treatment.
  Oxygenation index is the artery partial pressure of oxygen divided by the concentration of inhaled oxygen.

CONTACTS AND LOCATIONS:
Overall Officials: Zhongmin Liu, Dr., Study Chair — Shanghai East Hospital
Locations (1):
- Shanghai East Hospital, Shanghai Tongji University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No